CLINICAL TRIAL: NCT03059017
Title: Novel Nano-vesicles of Salbutamol Sulphate in Metered Dose Inhalers: Formulation, Characterization, In Vitro and In Vivo Evaluation
Brief Title: In Vivo Investigation of Novel Nano-vesicles of Salbutamol Sulphate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Mona Gamal Mohamed Afifi Arafa, Lecturer, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSMDI-2017-01
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Drug Effect; Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — Albuterol; Liposomes

STUDY DESIGN:
Intervention Model Description: Volunteers will be divided into two groups; each group contained 10 volunteers who will receive one formula of the selected formulae.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Niosomal salbutamol sulphate inhalers (Experimental): Niosomes
  Interventions: Drug: Niosomes
- salbutamol sulphate inhalers (Placebo Comparator): control testing
  Interventions: Drug: Salbutamol Sulphate

INTERVENTIONS:
Drug: Salbutamol Sulphate — salbutamol sulphate packaged as aerosol
  Arms: salbutamol sulphate inhalers
Drug: Niosomes — Niosomes
  Other Names: nano-vesicles
  Arms: Niosomal salbutamol sulphate inhalers

SUMMARY:
The relative bioavailability of different salbutamol sulphate inhaler formulations will be studied in healthy male subjects according to the ethical regulations of World Medical Association Declaration of Helsinki (1996) after the approval of the ethical committee, Faculty of Pharmacy, The British University in Egypt.

DETAILED DESCRIPTION:
In this study, 20 healthy, non smoking, adult male volunteers (age: 30-45 years, weight: 65-80 kg) will carry out screening procedures which include instruction and practice with the placebo metered dose inhaler devices that will be used in the study. In addition, all subjects were fully informed in writing of the objectives and implications of the trial. No subject will be considered for the study if developed any symptoms of allergic disorders. Subjects will follow a normal diet and will not receive any other medications. Volunteers will be divided into two groups; each group contained 10 volunteers who will receive one formula of the selected formulae.

Each volunteer will inhale eight puffs (4 puffs at -5 min & 4 puffs at 0 min) which are equivalent to 0.8 mg of salbutamol sulphate . To inhale through metered dose inhalers, volunteers will be trained to exhale slowly to their residual volume (as far as comfortable), put the inhaler into their mouth and seal their lips round the mouth piece. Then they will be instructed to take a slow deep inspiration to their total lung capacity over approximately 5-10 seconds. At the end of each inhalation, they will hold their breath for 10 seconds and then breathe normally (Ball et al, 2002) . Three milliliters of blood will be withdrawn at 0, 0.5, 1, 2, 3, 4, 5 and 6 h after administration. The blood will be heparinized immediately and centrifuged at 3000 rpm for 10 minutes. The plasma samples will be stored at freeze temperature until analysis. Two different formulae will be compared during the first six hours following administration. The maximum plasma concentration (Cmax), the time required to reach maximum plasma concentration (Tmax) and the area under plasma concentration time curve (AUC) will be calculated using validated Excel software.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Chronic disease
* Smoking
* Hospitalization

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2017-02-05 (Actual); Study Completion 2017-02-05 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | Twenty Four Hours
  The maximum concentration of Salbutamol Sulphate in human blood after time intervals 0, 30, 1,2, 3,4 , 5 & 6 hs will be calculated using validated using Excel software.

SECONDARY OUTCOMES:
The time required to reach maximum plasma (Tmax) | Twenty Four Hours
  Time taken for Salbutamol Sulphate to reach its maximum concentration in human blood & will be calculated using validated using Excel software

OTHER OUTCOMES:
The area under plasma concentration time curve (AUC) | Twenty Four Hours
  The integral in a plot of concentration of Salbutamol Sulphate in blood plasma against time.

IPD SHARING:
Plan to Share IPD: Yes
Share of the results by Publication

REFERENCES:
- [Background] Ball DJ, Hirst PH, Newman SP, Sonet B, Streel B, Vanderbist F. Deposition and pharmacokinetics of budesonide from the Miat Monodose inhaler, a simple dry powder device. Int J Pharm. 2002 Oct 1;245(1-2):123-32. doi: 10.1016/s0378-5173(02)00338-1. PMID 12270249
- [Background] Balanag VM, Yunus F, Yang PC, Jorup C. Efficacy and safety of budesonide/formoterol compared with salbutamol in the treatment of acute asthma. Pulm Pharmacol Ther. 2006;19(2):139-47. doi: 10.1016/j.pupt.2005.04.009. Epub 2005 Jul 11. PMID 16009588